CLINICAL TRIAL: NCT07238803
Title: Outcomes of Using Flexible and Navigable Suction Sheath With Flexible Ureteroscopy in Treatment of Lower Calyceal Stones: A Prospective Study
Brief Title: Outcomes of Using FANS With FURS in TTT of Lower Calyceal Stones.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mahmoud Ahmed Elsayed Ahmed Lasheen, Urology Resident, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 853
Record Dates: First submitted 2025-11-13; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Kidney Stone; Kidney Calculi
Keywords: Flexible Ureteroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main arm .. single arm (Experimental): Patients with lower calyceal stones
  Interventions: Device: flexible and navigable suction sheath with flexible ureteroscopy

INTERVENTIONS:
Device: flexible and navigable suction sheath with flexible ureteroscopy — placement of flexible and navigable suction sheath (FANS)which has an oblique side branch with pressure vent, that can be connected to negative pressure aspiration, and a flexible tip, allowing for efficient and effective treatment of urinary stones.
  * Flexible URS diameter will be at the least 2 Fr smaller than the sheath.
  * The main tube is closed by a rubber seal with a center aperture as the flexible ureteroscope pathway, The oblique tube with a pressure-regulating venting slit along the longitudinal axis acts as a suctioning channel connected to a vacuum device.
  * The inflow of irrigation is through the endoscope, the outflow of irrigation is between the scope and the sheath.
  * A vortex is created at the distal end of the sheath, the irrigation fluid, the stone fragments, dust, and blood, etc. in the vortex can be aspirated out.
  * The aspiration pressure can be adjusted by the pressure vent on the oblique side branch of the sheath.
  Other Names: FANS ureteral access sheath

SUMMARY:
The aim of this study is to evaluate and assess the outcomes of flexible ureteroscopy (FURS) with flexible and navigable suction UAS (FANS) in the treatment of lower calyceal stones.

DETAILED DESCRIPTION:
With the continued advancements of technology and increasing experience gained by urologists in ureteroscopic skills, fURS has become a standard treatment for kidney stones lesser than 2 cm in diameter. In the previous the European guidelines and American Urologic Association guidelines for management of urolithiasis, fURS were recommended as a second-line treatment for stones less than 2 cm after ESWL, however in the recent revision of the guidelines, RIRS can be used as the first-line management option especially for stones measuring between 11 and 20 mm.

The ureteral access sheath (UAS), initially introduced by Hisao Takayasu in 1974 Despite continued advances in retrograde intrarenal surgery (RIRS), recent real-world data for 6669 patients in the FLEXOR registry revealed residual fragments in 21.7% of patients, of whom 51.5% required a second intervention.

The sepsis rate in the same study was just 1.3%. Hence, there is still much to improve in terms of technical expertise and technology for RIRS. Many aids have been introduced to streamline RIRS and improve procedural success. These include suction via a scope or ureteral access sheath (UAS), postintervention catheters, slimmer single-use scopes, and high-power lasers, these improvements have made RIRS a standard of care according to international guidelines.

It has been reported that vacuum aided or suction aspiration sheaths have strong potential to improve the stone-free status (SFS) rate and minimize infectious compilations associated with the negative effects of high intrarenal pressure and temperature, However, the true potential of the advances for RIRS has yet to be investigated. The ideal game-changing technological innovation for RIRS should improve all key outcomes of the procedure, including the rate of immediate single stage SFS, perioperative and postoperative complications, and the reintervention rate for residual fragments. One recent advance that has shown much promise is a flexible and navigable sheath (FANS) So, we will conduct a prospective study to assess whether FANS could be a potential game-changer for RIRS in adults with lower calyceal stones instead of traditional UAS especially regarding stone-free rates (SFR), complications and cost.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years old.
2. Patients with lower calyceal stones scheduled for FURS.

Exclusion Criteria:

1. patients with active urinary tract infections.
2. Patients with renal and ureteric anomalies.
3. patients with coagulopathy
4. patients who are refusing to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Stone-Free Rate Following Flexible Ureteroscopy with FANS sheath for Management of Renal and Ureteral Calculi. | 1 month after the procedure (preferred and most common for SFR assessment)
  This clinical study aims to evaluate the stone-free rate (SFR) following flexible ureteroscopy (FURS) in patients with renal or ureteral calculi. The primary outcome measure is the proportion of patients who achieve complete stone clearance, as determined by postoperative imaging (non-contrast CT or ultrasound) within a defined follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Latif Mohammed Zayed, professor of urology, Study Director — Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon reasonable request from qualified researchers after study completion. A data dictionary will also be provided.
  Time Frame: 6 months after final publication, available for 3 years. Access Criteria: Contact the principal investigator.